CLINICAL TRIAL: NCT07117097
Title: Minimally Invasive Non- Surgical Periodontal Therapy of Intrabony Defects: Molecular Healing Patterns and the Impact of Smoking on Outcomes
Brief Title: Minimally Invasive Non- Surgical Periodontal Therapy of Intrabony Defects: Healing Patterns and Smoking Impact
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: 251 Hellenic Air Force & VA General Hospital (Other)
Responsible Party: Principal Investigator, ILIAS OIKONOMOU, Principal Investigator, Periodontist, Department of Periodontology, 251 Hellenic Air Force & VA Hospital, Athens, Greece, Doctoral researcher, Department of Periodontology, Institute of Dentistry, University of Turku, Turku, Finland, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Φ076/13310/Σ6276/5Νοε24/251ΓΝΑ
Record Dates: First submitted 2025-03-31; First posted 2025-08-12 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Periodontitis
Keywords: Periodontitis; Intrabony defect; GCF; Minimally invasive; smoking; non surgical; bone
MeSH Terms: conditions — Periodontitis; Smoking | interventions — Tooth Exfoliation; Root Planing; Periodontal Debridement

STUDY DESIGN:
Intervention Model Description: At first a Randomized Controlled clinical trial study (RCT) will be conducted and then a prospective cohort study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Non-smokers cNSPT (Active Comparator): Participants will be non-smokers. Periodontal treatment intervention will include: thorough debridement of the root surface under local anaesthesia, using conventional piezoelectric devices (EMS, Switzerland) and hand instruments (Gracey, Hu Friedy).
  Interventions: Procedure: conventional Non-Surgical Periodontal Treatment (cNSPT)
- Non-smokers MINST (Experimental): Participants will be non-smokers. Periodontal treatment intervention will include: local anaesthesia by infiltration without adrenaline, thorough debridement of the root surface through a subpapillary access using exclusively piezoelectric devices with specific thin and delicate tips (EMS, Switzerland) and 4X magnification loupes, taking care to minimize the soft tissue trauma and to stimulate the formation of a stable blood clot.
  Interventions: Procedure: Minimally Invasive Non- Surgical Periodontal Therapy (MINST)
- Smokers MINST (Experimental): Participants will be smokers. Periodontal treatment intervention will include: local anaesthesia by infiltration without adrenaline, thorough debridement of the root surface through a subpapillary access using exclusively piezoelectric devices with specific thin and delicate tips (EMS, Switzerland) and 4X magnification loupes, taking care to minimize the soft tissue trauma and to stimulate the formation of a stable blood clot.
  Interventions: Procedure: Minimally Invasive Non- Surgical Periodontal Therapy (MINST)

INTERVENTIONS:
Procedure: Minimally Invasive Non- Surgical Periodontal Therapy (MINST) — The procedure consists of thorough debridement of the root surface through a subpapillary access using exclusively piezoelectric devices with specific thin and delicate tips (EMS, Switzerland) and 4X magnification loupes, taking care to minimize the soft tissue trauma and to stimulate the formation of a stable blood clot
  Arms: Non-smokers MINST; Smokers MINST
Procedure: conventional Non-Surgical Periodontal Treatment (cNSPT) — The intervention consists of thorough debridement of the root surface under local anaesthesia, using conventional piezoelectric devices and hand instruments
  Other Names: scaling and root planing; SRP; non-surgical periodontal treatment; periodontal debridement
  Arms: Non-smokers cNSPT

SUMMARY:
This study is consisted of two arms. At first, a randomized controlled clinical trial will be conducted. Eighty systematically healthy, non-smoker patients with Periodontitis stage III or IV, grades B to C will be included. Each patient will have to present one intrabony defect site ( site with Probing Depth (PD)>5mm and radiographic defect depth > or =3mm). The patients will be randomized in two groups, regarding the treatment intervention of the intrabony defects: Group A (conventional Non-Surgical Periodontal Treatment, cNSPT) and Group B (Minimally Invasive Non-Surgical Therapy, MINST). At 5 days and 3 months following intervention, GCF samples will be collected from the intrabony defects in order to assess the molecular healing patterns through intergroup comparisons of inflammation and healing biomarkers. Then two prospective cohort studies will be conducted. The Group B patients will be matched with forty systematically healthy, smoker patients (Group C) with Periodontitis stage III or IV, grades B to C with each one presenting one intrabony defect site ( site with Probing Depth (PD)>5mm and radiographic defect depth > or =3mm). Then MINST will be performed in the patients of Group C and the two groups will be compared regarding the clinical and radiographic data obtained by clinical and radiographic examinations performed in both groups' intrabony defects pre-treatment and 6 months following the intervention (first prospective study) and regarding the differences in regeneration biomarkers in GCF samples obtained from the intrabony defects 5 days and 3 months post-treatment (second prospective study).

DETAILED DESCRIPTION:
The aim of this study is to define the possible differences of molecular healing response between MINST and cNSPT and, also, between smokers and non-smokers after MINST and to examine whether smoking is associated with inferior clinical outcomes after MINST.

The specific objectives of our study are:

1. To compare the response of non-smokers after MINST and cNSPT in terms of inflammation and healing GCF biomarkers,
2. To compare the response of non-smokers and smokers after MINST, in terms of clinical and radiographic outcomes,
3. To compare the response of non-smokers and smokers after MINST, in terms of regeneration GCF biomarkers.

3. Research implementation

1. Randomized controlled clinical trial (RCT) study

   A statistical power analysis program (GPower 3.1, Franz Faul, Universität Kiel, Kiel, Germany) was used for the sample size calculation. Since there were no prior studies comparing MINST and cNSPT in terms of their GCF biomarker levels, the effect size was be defined based on previous research reporting significantly different gingival crevicular fluid levels of biomarkers between periodontitis and health. Firstly a parallel-group, single centre, examiner-blind randomized controlled trial will be conducted. Eighty systematically healthy, non-smoker patients with Periodontitis stage III or IV, grades B to C will be included. Each patient will have to present one intrabony defect site ( site with Probing Depth (PD)>5mm and radiographic defect depth > or =3mm). The patients will be randomized into one of the following periodontal treatment modality groups regarding the intrabony defect:
   * Group A: cNSPT
   * Group B: MINST The patients will receive periodontal cause related therapy, including comprehensive oral hygiene instructions and full- mouth conventional NSPT, namely Phase I therapy with piezoelectric devices (EMS, Switzerland) and hand instruments (Gracey, Hu Friedy) under local anaesthesia. Specifically in the intrabony defects included, the intervention will be performed according to each patient's group allocation.

   At 5 days and 3 months following intervention, GCF samples will be collected from the intrabony defects in order to assess the molecular healing patterns through intergroup comparisons of inflammation and healing biomarkers.
2. Prospective cohort studies Subsequently patients of Group B will be matched with forty smoker patients with Periodontitis stage III or IV, grades B to C for age and sex, with each of them presenting one intrabony defect site ( site with Probing Depth (PD)>5mm and radiographic defect depth > or =3mm). These patients (Group C) will receive the same full-mouth periodontal treatment management as Groups A and B and regarding the intrabony defects included, MINST interventions will be performed.

   A prospective cohort study will be conducted to assess the differences in treatment outcomes after MINST in smokers and in non-smokers, by comparing clinical and radiographic data obtained by clinical and radiographic examinations performed in both groups' intrabony defects pre-treatment and 6 months following the intervention.

   Also, a prospective cohort study will be conducted to compare the molecular healing patterns in smokers and non-smokers after MINST, via assessment of the differences in regeneration biomarkers in GCF samples obtained from the intrabony defects 5 days and 3 months post-treatment.
3. Participants All patients who will be included in the study will be periodontal patients seeking treatment at the Department of Periodontology, 251 Hellenic Airforce General Hospital, Athens, Greece.

   All participants should be free of any systemic or oral conditions that could affect disease progression or treatment outcomes. Thus reasons for exclusion will be: medical history including diabetes, hepatic or renal disease, history of conditions requiring prophylactic antibiotics, anti-inflammatory or anticoagulant therapy the preceding month, systemic antibiotic therapy the preceding 3 months, history of alcohol or drug abuse, self-reported pregnancy or lactation, other severe acute or chronic medical or psychiatric condition, periodontal treatment within the last 12 months and presence of drug-induced gingival overgrowth. As smokers will be defined patients who are current smokers and smoke at least 10 cigarettes per day. As non-smokers will be considered patients who have never smoked or who have quit smoking for 5 years at least.
4. Ethical Considerations These studies will be conducted in full accordance with the guidelines of the Declaration of Helsinki. Ethical approval will be requested from the Ethics and Research Committee of the 251 Hellenic Airforce General Hospital, Athens, Greece (date of application 09/2024).
5. Clinical Intra-oral Examination Plaque index (PI), gingival index (GI), bleeding on probing (BoP), probing depth (PD), gingival recession (REC) and clinical attachment level (CAL) will be recorded at the involved tooth site and also full mouth to establish a diagnosis by a single-blinded, calibrated examiner, using a computerized pressure sensitive probe (Florida Probe).
6. Radiographic examination Periapical digital radiographs will be taken using the parallel cone technique with a customized radiographic stent. Radiographic measurements will be made using a software programme (ImageJ, Oracle Corporation, San Jose, California) by a single-blinded, calibrated examiner and will include: the distance between the tooth cementoenamel junction (CEJ) and the bottom of the intrabony defect, the distance between the CEJ and the alveolar bone crest, the depth of the intrabony defect and the angle of the intrabony defect (defined by the lines of the tooth root surface and the defect's bone wall)21.
7. GCF Collection and analysis GCF sampling will be performed for 30s using Periopaper (OraFlow Inc., New York) placed at the entrance of the sulcus. Volumes of GCF samples will be determined with a Periotron (OraFlow Inc., New York) device immediately after the sample collection. Afterwards, the samples will be stored dry in Eppendorf tubes at -80°C s until the day of analyze. At the day of analyze, GCF will be eluted in 200μl of PBS (with 0.1% BSA). Biomarker levels in GCF samples will be determined by Luminex method using commercial kits.
8. MINST and cNSPT treatment interventions in the intrabony defects MINST treatment protocol will include: local anaesthesia by infiltration without adrenaline, thorough debridement of the root surface through a subpapillary access using exclusively piezoelectric devices with specific thin and delicate tips (EMS, Switzerland) and 4X magnification loupes, taking care to minimize the soft tissue trauma and to stimulate the formation of a stable blood clot22.

   cNSPT treatment protocol will include thorough debridement of the root surface under local anaesthesia, using conventional piezoelectric devices (EMS, Switzerland) and hand instruments (Gracey, Hu Friedy).
9. Statistical analysis Following the detection of the data distribution with the Kolmogorov-Smirnov test, repeated t-test or ANOVA in case of normal distribution will be used in the statistical analysis, and the Mann-Whitney U or Kruskal Wallis tests in case of non-normal distribution. Repeated Measures ANOVA and Linear Mixed Models will be used to compare parameters between visits. In determining the correlation between chemokine concentrations and clinical parameters, the parametric Pearson test or the non-parametric Spearman test will be used according to the distribution.

ELIGIBILITY:
Inclusion Criteria:

* patients with Periodontitis stage III or IV, grades B to C . Each patient will have to present one intrabony defect site ( site with Probing Depth (PD)>5mm and radiographic defect depth >3mm).
* participants should be free of any systemic or oral conditions that could affect disease progression or treatment outcomes

Exclusion Criteria:

* diabetes
* hepatic or renal disease
* history of conditions requiring prophylactic antibiotics
* anti-inflammatory or anticoagulant therapy the preceding month
* systemic antibiotic therapy the preceding 3 months
* history of alcohol or drug abuse
* self-reported pregnancy or lactation
* other severe acute or chronic medical or psychiatric condition
* periodontal treatment within the last 12 months
* presence of drug-induced gingival overgrowth

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Concentrations of GCF inflammation and regeneration biomarkers. | At 5 days and 3 months following intervention
  Concentrations will be measured in pg/ml
Total amounts of GCF inflammation and regeneration biomarkers | At 5 days and 3 months following intervention
  Total amounts will be measured in pg/30 s

SECONDARY OUTCOMES:
Plaque index (PI) | pre-treatment and 6 months following the intervention
  Recorded in a dichotomous manner (+ or -) using a UNC-15 periodontal probe
Gingival index (GI) | pre-treatment and 6 months following the intervention
  Recorded in a dichotomous manner (+ or -) using a UNC-15 periodontal probe
Bleeding on probing (BoP) | pre-treatment and 6 months following the intervention
  Recorded in a dichotomous manner (+ or -) using a UNC-15 periodontal probe
Probing depth (PD) | pre-treatment and 6 months following the intervention
  Measured in mm using a UNC-15 periodontal probe
Gingival recession (REC) | pre-treatment and 6 months following the intervention
  Measured in mm using a UNC-15 periodontal probe
Clinical attachment level (CAL) | pre-treatment and 6 months following the intervention
  Measured in mm using a UNC-15 periodontal probe
Distance between the tooth cementoenamel junction (CEJ) and the bottom of the intrabony defect | pre-treatment and 6 months following the intervention
  Radiographic measurement in mm
Distance between the CEJ and the alveolar bone crest | pre-treatment and 6 months following the intervention
  Radiographic measurement in mm
Depth of the intrabony defect | pre-treatment and 6 months following the intervention
  Radiographic measurement in mm
Angle of the intrabony defect | pre-treatment and 6 months following the intervention
  Radiographic measurement in degrees

CONTACTS AND LOCATIONS:
Overall Officials: ILIAS OIKONOMOU, DDS,MSc, Principal Investigator — Institute of Dentistry, University of Turku, Turku, Finland; Ulvi Gürsoy, DDS, PhD, Study Director — Institute of Dentistry, University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared upon request. Data will be made available only after a structured proposal is submitted, reviewed, and approved by the study team. Access will be granted for research purposes that align with the study objectives, and data will be shared through a secure platform upon signing a data use agreement.
Access Criteria: The IPD sharing requests will be reviewed by the principal investigator and the study director.

REFERENCES:
- [Background] Nibali L, Koidou V, Salomone S, Hamborg T, Allaker R, Ezra R, Zou L, Tsakos G, Gkranias N, Donos N. Minimally invasive non-surgical vs. surgical approach for periodontal intrabony defects: a randomised controlled trial. Trials. 2019 Jul 27;20(1):461. doi: 10.1186/s13063-019-3544-8. PMID 31351492
- [Background] Anoixiadou S, Parashis A, Vouros I. Enamel matrix derivative as an adjunct to minimally invasive non-surgical treatment of intrabony defects: A randomized clinical trial. J Clin Periodontol. 2022 Feb;49(2):134-143. doi: 10.1111/jcpe.13567. Epub 2021 Nov 9. PMID 34708441
- [Background] Reynolds MA, Kao RT, Camargo PM, Caton JG, Clem DS, Fiorellini JP, Geisinger ML, Mills MP, Nares S, Nevins ML. Periodontal regeneration - intrabony defects: a consensus report from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S105-7. doi: 10.1902/jop.2015.140378. Epub 2014 Oct 15. PMID 25315019
- [Background] Kotsakis GA, Javed F, Hinrichs JE, Karoussis IK, Romanos GE. Impact of cigarette smoking on clinical outcomes of periodontal flap surgical procedures: a systematic review and meta-analysis. J Periodontol. 2015 Feb;86(2):254-63. doi: 10.1902/jop.2014.140452. Epub 2014 Oct 9. PMID 25299388
- [Background] Chang J, Meng HW, Lalla E, Lee CT. The impact of smoking on non-surgical periodontal therapy: A systematic review and meta-analysis. J Clin Periodontol. 2021 Jan;48(1):60-75. doi: 10.1111/jcpe.13384. Epub 2020 Nov 5. PMID 33022758
- [Background] Haber J, Wattles J, Crowley M, Mandell R, Joshipura K, Kent RL. Evidence for cigarette smoking as a major risk factor for periodontitis. J Periodontol. 1993 Jan;64(1):16-23. doi: 10.1902/jop.1993.64.1.16. PMID 8426285
- [Background] Liu S, Hu B, Zhang Y, Li W, Song J. Minimally Invasive Surgery Combined with Regenerative Biomaterials in Treating Intra-Bony Defects: A Meta-Analysis. PLoS One. 2016 Jan 19;11(1):e0147001. doi: 10.1371/journal.pone.0147001. eCollection 2016. PMID 26785405
- [Background] Mehta J, Montevecchi M, Garcia-Sanchez R, Onabolu O, Linares A, Eriksson F, Ghezzi C, Donghi C, Lu EM, Nibali L. Minimally invasive non-surgical periodontal therapy of intrabony defects: A prospective multi-centre cohort study. J Clin Periodontol. 2024 Jul;51(7):905-914. doi: 10.1111/jcpe.13984. Epub 2024 May 6. PMID 38710583
- [Background] Nibali L, Yeh YC, Pometti D, Tu YK. Long-term stability of intrabony defects treated with minimally invasive non-surgical therapy. J Clin Periodontol. 2018 Dec;45(12):1458-1464. doi: 10.1111/jcpe.13021. Epub 2018 Nov 5. PMID 30307641
- [Background] Nibali L, Pometti D, Chen TT, Tu YK. Minimally invasive non-surgical approach for the treatment of periodontal intrabony defects: a retrospective analysis. J Clin Periodontol. 2015 Sep;42(9):853-859. doi: 10.1111/jcpe.12443. Epub 2015 Sep 29. PMID 26257238
- [Background] Cortellini P, Tonetti MS. Clinical and radiographic outcomes of the modified minimally invasive surgical technique with and without regenerative materials: a randomized-controlled trial in intra-bony defects. J Clin Periodontol. 2011 Apr;38(4):365-73. doi: 10.1111/j.1600-051X.2011.01705.x. Epub 2011 Feb 8. PMID 21303402
- [Background] Koop R, Merheb J, Quirynen M. Periodontal regeneration with enamel matrix derivative in reconstructive periodontal therapy: a systematic review. J Periodontol. 2012 Jun;83(6):707-20. doi: 10.1902/jop.2011.110266. Epub 2011 Nov 3. PMID 22050544
- [Background] Cortellini P, Tonetti MS. Improved wound stability with a modified minimally invasive surgical technique in the regenerative treatment of isolated interdental intrabony defects. J Clin Periodontol. 2009 Feb;36(2):157-63. doi: 10.1111/j.1600-051X.2008.01352.x. PMID 19207892
- [Background] Cortellini P, Tonetti MS. A minimally invasive surgical technique with an enamel matrix derivative in the regenerative treatment of intra-bony defects: a novel approach to limit morbidity. J Clin Periodontol. 2007 Jan;34(1):87-93. doi: 10.1111/j.1600-051X.2006.01020.x. PMID 17243998
- [Background] Rams TE, Listgarten MA, Slots J. Radiographic alveolar bone morphology and progressive periodontitis. J Periodontol. 2018 Apr;89(4):424-430. doi: 10.1002/JPER.17-0279. PMID 29683496
- [Background] Nibali L, Koidou VP, Nieri M, Barbato L, Pagliaro U, Cairo F. Regenerative surgery versus access flap for the treatment of intra-bony periodontal defects: A systematic review and meta-analysis. J Clin Periodontol. 2020 Jul;47 Suppl 22:320-351. doi: 10.1111/jcpe.13237. PMID 31860134
- [Background] Lang NP. Focus on intrabony defects--conservative therapy. Periodontol 2000. 2000 Feb;22:51-8. doi: 10.1034/j.1600-0757.2000.2220105.x. No abstract available. PMID 11276516
- [Background] Graziani F, Karapetsa D, Alonso B, Herrera D. Nonsurgical and surgical treatment of periodontitis: how many options for one disease? Periodontol 2000. 2017 Oct;75(1):152-188. doi: 10.1111/prd.12201. PMID 28758300
- [Background] Tonetti MS, Jepsen S, Jin L, Otomo-Corgel J. Impact of the global burden of periodontal diseases on health, nutrition and wellbeing of mankind: A call for global action. J Clin Periodontol. 2017 May;44(5):456-462. doi: 10.1111/jcpe.12732. Epub 2017 May 8. PMID 28419559
- [Background] Kassebaum NJ, Bernabe E, Dahiya M, Bhandari B, Murray CJ, Marcenes W. Global burden of severe periodontitis in 1990-2010: a systematic review and meta-regression. J Dent Res. 2014 Nov;93(11):1045-53. doi: 10.1177/0022034514552491. Epub 2014 Sep 26. PMID 25261053
- [Background] Corbella S, Calciolari E, Alberti A, Donos N, Francetti L. Systematic review and meta-analysis on the adjunctive use of host immune modulators in non-surgical periodontal treatment in healthy and systemically compromised patients. Sci Rep. 2021 Jun 9;11(1):12125. doi: 10.1038/s41598-021-91506-7. PMID 34108528